CLINICAL TRIAL: NCT05594836
Title: The Effect of Infant Calming Training Given to Primiparous Mothers on Perception of Maternal Role, Maternal Attachment and Breastfeeding Self-Efficacy
Brief Title: The Effect of Infant Calming Education on Maternal Role Perception, Maternal Attachment and Breastfeeding Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/692
Record Dates: First submitted 2022-10-20; First posted 2022-10-26 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Infant Development

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Perception of Maternal Role, Maternal Attachment and Breastfeeding Self-Efficacy
  Interventions: Behavioral: Infant Calming Training
- control (No Intervention): not Perception of Maternal Role, Maternal Attachment and Breastfeeding Self-Efficacy

INTERVENTIONS:
Behavioral: Infant Calming Training — Perception of Maternal Role, Maternal Attachment and Breastfeeding Self-Efficacy during Infant Calming Training
  Arms: Training

SUMMARY:
The research is a randomized controlled experimental study. The study includes primiparous mothers hospitalized in the Obstetrics and Gynecology Service of Recep Tayyip Erdogan University Training and Research Hospital between 01/12/2022-01/10/2023.

The population of the study will be composed of primiparous mothers hospitalized in the Obstetrics and Gynecology Service of Recep Tayyip Erdoğan University Training and Research Hospital between 01/12/2022 and 01/10/2023. All mothers who were hospitalized in the gynecology service during the data collection period and met the inclusion criteria will be included in the study and sample selection will not be made.

"Mother and Baby Descriptive Information Form", "Maternal Attachment Scale", "Postpartum Breastfeeding Self-Efficacy Scale-Short Form", "Semantic Difference Scale-Me as Mother" and "Sleep and Crying Diary" will be used to collect research data. Developing the 5S application, which is a baby calming technique, as an educational material in the research. A training booklet will be prepared and used by making use of the training materials that Harvey Karp shared with the researchers.

DETAILED DESCRIPTION:
Type of Research The research is a randomized controlled experimental study. Place and Time of the Research The study includes primiparous mothers hospitalized in the Obstetrics and Gynecology Service of Recep Tayyip Erdogan University Training and Research Hospital between 01/12/2022-01/10/2023.

Population and Sample of the Research The population of the study will be composed of primiparous mothers hospitalized in the Obstetrics and Gynecology Service of Recep Tayyip Erdoğan University Training and Research Hospital between 01/12/2022 and 01/10/2023. All mothers who were hospitalized in the gynecology service during the data collection period and met the inclusion criteria will be included in the study and sample selection will not be made.

Data Collection Tools "Mother and Baby Descriptive Information Form", "Maternal Attachment Scale", "Postpartum Breastfeeding Self-Efficacy Scale-Short Form", "Semantic Difference Scale-Me as Mother" and "Sleep and Crying Diary" will be used to collect research data. Developing the 5S application, which is a baby calming technique, as an educational material in the research. A training booklet will be prepared and used by making use of the training materials that Harvey Karp shared with the researchers.

Data Collection The mothers in the control and education groups who meet the inclusion criteria of the study will be verbally informed about the purpose of the study and the method of application. "Informed Consent Form" will be filled in for mothers who agree to participate in the study. Data collection will not be carried out simultaneously with the mothers in the training and control groups, in case the mothers in the ward may be affected by the training provided. According to a computer-generated randomization list, patients will be assigned to one of two groups using the closed-envelope technique.

Control Group: Mothers in the control group will not be given any treatment other than the standard neonatal care routinely given in the clinic. Mother and Baby Descriptive Information Form, Semantic Difference Scale (Me as a Mother) and Breastfeeding Self-Efficacy Scale will be filled in by face-to-face interview method, and the Baby Sleep Descriptive Information Form will be filled in during a period of time when the baby is sleeping and the mother is feeling well. and how to fill out the Crying Diary. Since it was deemed appropriate to collect the maternal attachment scale in the first and fourth months after birth, the data of the Maternal Attachment Scale will be collected via the online questionnaire sent to the mothers at the 4th week after birth. At the end of the 8th week, the data will be filled again with the Semantic Difference Scale (Me as the Mother), Maternal Attachment and Breastfeeding Self-Efficacy Scale from the mothers. Baby Sleep and Crying Diary forms will be received.

Training Group: Primiparous mothers followed in the gynecology service in the postpartum period will be given face-to-face Infant Calming Training, which lasts for approximately 30 minutes, during a time when the baby is sleeping and the mother is feeling well. After the training, the Mother and Baby Introductory Information Form, the Semantic Difference Scale (Me as the Mother) and the Breastfeeding Self-Efficacy Scale will be filled in by face-to-face interview method and information will be given on how to fill the Baby Sleep and Crying Diary. The mother will be given a blanket to swaddle her baby along with the prepared educational material, and the Sleeping Companion with a White Noise Sensor will be given to the mother. The data of the Maternal Attachment Scale will be collected through the online questionnaire sent to the mothers in the 4th week after birth. Meaning from mothers at the end of the 8th week. Data will be replenished with the Salary Difference Scale (Me as a Mother), Maternal Attachment and Breastfeeding Self-Efficacy Scale. Baby Sleep and Crying Diary forms will be received.

Evaluation of Data Evaluation of statistics will be done by blinding method. The analysis of the data will be done by the statistician. After ensuring that the data is coded and labeled in a way that preserves the blinding, the data will be submitted and data analysis will be performed.

The data will be analyzed with the SPSS for Windows 22 package program. The normality distribution of the data will be determined by the Kurtosis and Skewness coefficients. In the analysis of the data, numbers, percentages, mean and standard deviations, as well as the t-test for normally distributed measurements in the comparison of paired groups, for independent groups, and Mann Whitney U analysis for non-normally distributed measurements will be used. In the comparison of multiple groups, analysis of variance will be used for normally distributed measurements. Statistical significance will be accepted as p<0.05.

Ethical Principles of Research In order to carry out the research, official permission will be obtained from the relevant institution with ethical approval from the Ethics Committee of Atatürk University Faculty of Medicine. The purpose of the study will be explained to the mothers who meet the research group criteria, their questions will be answered and their verbal and written consents will be obtained. The mothers will be informed that the data collected during the research will be processed anonymously, confidentially, and will not be used outside of the study in question, and that they can leave the study whenever they wish. Since the research is based on the use of data obtained from humans, and therefore, due to the necessity of observing personal rights, the relevant ethical principles "Informed Consent", "Volunteerism" and "Protection of Confidentiality" will be followed.

ELIGIBILITY:
Inclusion Criteria:

Maternal criteria;

* Being primiparous
* Being over 18 years old
* Being literate
* Absence of multiple pregnancy
* Volunteering to participate in the research
* Being open to communication and interaction
* Owning a smartphone (for education group - white noise) Criteria for the baby;
* Being older than 37 weeks of gestation
* Normal birth weight (between 2500-4000 g)
* Absence of a medical condition that would prevent sucking

Exclusion Criteria:

* Admission of the baby to the intensive care unit
* The presence of a chronic disease in the mother that will prevent baby care
* Having any diagnosed disease of the baby during the study
* Artificial feeding of the baby

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Maternal Attachment Scale | 9 MONTHS
  The highest level of attachment occurs when the mother understands the baby's signs and symptoms and meets the baby's physical and emotional needs. A mother's loving attachment to her baby, that is, maternal attachment, is one of the most important elements that promotes the healthy growth and development of the child.
  MBI was developed in 1994. MDS is a 4-point Likert-type scale that includes 26 items and is answered between always (4 points) and never (1 point). An overall score is obtained from the sum of all items. The lowest score that can be obtained from the scale is 26, and the highest score is 104. A high score indicates high maternal attachment. The validity and reliability of the scale for Turkish society was carried out in 2009 and it was determined that it would be suitable for mothers who have babies between one and four months after birth.
Postpartum Breastfeeding Self-Efficacy Scale-Short Form | 9 MONTHS
  It was developed in 1999 to evaluate mothers' breastfeeding self-efficacy levels. The first version of the scale consists of 33 items. Later, in 2003, a 14-item short form of the scale was developed. It is easier to apply and evaluates self-efficacy correctly. The Breastfeeding Self-Efficacy Short Form is a five-point Likert-type scale (1= "I am not sure at all" and 5 = "I am always sure"). The minimum score that can be obtained from the scale is 14, and the maximum score is 70. The higher the score, the higher the breastfeeding self-efficacy. The Turkish validity and reliability study of the scale was carried out in 2010.
Semantic Difference Scale-Me as Mother | 9 MONTHS
  This scale measures the evaluation dimensions of the concept of "myself as a mother". The scale consists of 11 semantic pairs of opposite adjectives with 11 items and 7 points. These 11 items are distributed within the 22 item opposite adjective pairs in the scale. Three items were evaluated with reverse scoring to prevent the participant from being biased while responding. The third, seventh, and eighth items were evaluated over "one" point instead of "seven" point. High total scores indicate positive maternal self-assessment. The scale was adapted to Turkish society in 2003.

CONTACTS AND LOCATIONS:
Overall Officials: ARZU SARIALİOĞLU, PHD, Study Director — Ataturk University
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED